CLINICAL TRIAL: NCT06010953
Title: An Open-label and Multicenter Phase Ib/II Clinical Trial to Evaluate the Safety, Immunogenicity, PK/PD Profile of SS109 and NovoSeven® Following a Single Dose, and the Preliminary Efficacy and Safety of SS109 During On-demand Treatment in Hemophilia Patients With Coagulation Factor VIII or IX Inhibitors
Brief Title: SS109 and NovoSeven ® PK / PD Profile, and Preliminary Efficacy and Safety of SS109 on Demand Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-109-I02
Record Dates: First submitted 2023-08-15; First posted 2023-08-25 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-11

CONDITIONS: Male; Hemophilia A With Inhibitor; Hemophilia B With Inhibitor; Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PK period: Cohort 1 (90 μg/kg) and Cohort 2 (270 μg/kg) (Experimental): In the PK study period, subjects are divided into 2 cohorts (90 μg/kg and 270 μg/kg), which are sequentially conducted. Cohort 1 (90 μg/kg) enrollment is performed firstly, and Cohort 2 (270 μg/kg) enrollment is performed after Cohort 1 enrollment is completed. Subjects enter the PK study period as non-randomized. All screened eligible subjects will receive a single dose of comparator NovoSeven® in the absence of significant active hemorrhage, followed by PK/PD sample collection; then receive a single dose of the same dose of investigational drug SS109, followed by PK/PD sample collection.
  Interventions: Drug: SS109
- On-demand treatment period: Group 1：90 μg/kg Group 2：180 μg/kg Group 3：270 μg/kg (Experimental): After completion of the PK study period, subjects will enter a 90-day on-demand treatment period and will be randomized into 3 groups (Group 1: 90 µg/kg, Group 2: 180 µg/kg, and Group 3: 270 µg/kg) at a ratio of 1:1:1. During on-demand treatment, subjects are treated on-demand with SS109 at the time of a new hemorrhage event and their efficacy is observed.
  Interventions: Drug: SS109

INTERVENTIONS:
Drug: SS109 — on-demand treatment with SS109 at the time of a new hemorrhage event

SUMMARY:
This is an open-label, multicenter Phase 1Ib/2II clinical trial of SS109 in adult hemophilia patients (≥ 18 years) with FVIII or FIX inhibitors to evaluate the PK/PD profile of SS109 and NovoSeven® after a single dose in adult hemophilia patients with FVIII or FIX inhibitors, to assess the preliminary efficacy and PK profile of SS109 during on-demand treatment, and to observe the safety and immunogenicity of SS109 throughout the study.

The trial consists of three periods: screening period, PK study period, and on-demand treatment period.

In the PK study period, subjects are divided into 2 cohorts (90 μg/kg and 270 μg/kg), which are sequentially conducted. Cohort 1 (90 μg/kg) enrollment is performed firstly, and Cohort 2 (270 μg/kg) enrollment is performed after Cohort 1 enrollment is completed. Subjects enter the PK study period as non-randomized. All screened eligible subjects will receive a single dose of comparator NovoSeven® in the absence of significant active hemorrhage, followed by PK/PD sample collection; then receive a single dose of the same dose of investigational drug SS109, followed by PK/PD sample collection. Specific times for PK/PD sample collection are listed in the schedule for biological sample collection.

After completion of the PK study period, subjects will enter a 90-day on-demand treatment period and will be randomized into 3 groups (Group 1: 90 µg/kg, Group 2: 180 µg/kg, and Group 3: 270 µg/kg) at a ratio of 1:1:1. During on-demand treatment, subjects are treated on-demand with SS109 at the time of a new hemorrhage event and their efficacy is observed. The investigator will judge the severity of subject's hemorrhage according to the type, location, clinical symptoms and signs of the subject's hemorrhage. Appropriate hemostatic treatment regimens and whether or not to perform the first SS109 on-demand treatment for the hemorrhage event at home may be developed by the investigator based on the subject's on-demand treatment group, according to the severity of hemorrhage and the recommended dosing frequency of SS109 (see Dosage/Regimen), and the dosing interval may be adjusted in conjunction with the subject's response to treatment. If the subject's last hemostatic treatment is administered within one week before the D96 visit point during the on-demand treatment period, the subject is required to continue follow-up observation for one week after the last dose before completing the end of study visit. PK/PD samples will be collected as appropriate during on-demand treatment, as specified in the schedule for biological sample collection.Observe subject safety throughout the study.

DETAILED DESCRIPTION:
This is an open-label, multicenter Phase 1Ib/2II clinical trial of SS109 in adult hemophilia patients (≥ 18 years) with FVIII or FIX inhibitors to evaluate the PK/PD profile of SS109 and NovoSeven® after a single dose in adult hemophilia patients with FVIII or FIX inhibitors, to assess the preliminary efficacy and PK profile of SS109 during on-demand treatment, and to observe the safety and immunogenicity of SS109 throughout the study.

The trial consists of three periods: screening period, PK study period, and on-demand treatment period.

In the PK study period, subjects are divided into 2 cohorts (90 μg/kg and 270 μg/kg), which are sequentially conducted. Cohort 1 (90 μg/kg) enrollment is performed firstly, and Cohort 2 (270 μg/kg) enrollment is performed after Cohort 1 enrollment is completed. Subjects enter the PK study period as non-randomized. All screened eligible subjects will receive a single dose of comparator NovoSeven® in the absence of significant active hemorrhage, followed by PK/PD sample collection; then receive a single dose of the same dose of investigational drug SS109, followed by PK/PD sample collection. Specific times for PK/PD sample collection are listed in the schedule for biological sample collection.

After completion of the PK study period, subjects will enter a 90-day on-demand treatment period and will be randomized into 3 groups (Group 1: 90 µg/kg, Group 2: 180 µg/kg, and Group 3: 270 µg/kg) at a ratio of 1:1:1. During on-demand treatment, subjects are treated on-demand with SS109 at the time of a new hemorrhage event and their efficacy is observed. The investigator will judge the severity of subject's hemorrhage according to the type, location, clinical symptoms and signs of the subject's hemorrhage. Appropriate hemostatic treatment regimens and whether or not to perform the first SS109 on-demand treatment for the hemorrhage event at home may be developed by the investigator based on the subject's on-demand treatment group, according to the severity of hemorrhage and the recommended dosing frequency of SS109 (see Dosage/Regimen), and the dosing interval may be adjusted in conjunction with the subject's response to treatment. If the subject's last hemostatic treatment is administered within one week before the D96 visit point during the on-demand treatment period, the subject is required to continue follow-up observation for one week after the last dose before completing the end of study visit. PK/PD samples will be collected as appropriate during on-demand treatment, as specified in the schedule for biological sample collection.

Observe subject safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years at the time of informed consent, male;
2. Patients with clinical diagnosis of hemophilia A or B (FVIII activity level ≤ 1% or FIX activity level ≤ 2% in the previous or screening period) who meet one of the following conditions:

   FVIII or FIX inhibitor level ≥ 5 Bu/mL at screening; FVIII or FIX inhibitor level < 5 Bu/mL and ≥ 0.6 Bu/mL at screening, with a high response to coagulation factor VIII or IX for injection (i.e., the patient has a previous history of positive FVIII/FIX inhibitor and inhibitor levels are ≥ 5 Bu/mL after reinfusion of FVIII/FIX).
3. No active bleeding symptoms prior to the first dose;
4. Subjects or impartial witnesses fully understand and comply with the requirements of the study protocol and are willing to complete the study as planned, and voluntarily cooperate in providing biological samples for testing as required by the protocol;
5. Be able to understand the procedures and methods of this clinical trial, and after fully informed consent, the patient voluntarily participates and signs the informed consent form by the patient himself or an impartial witness.

Exclusion Criteria:

1. Patients with a known history of hypersensitivity to the investigational product or any of its components;
2. Patients with previous hypersensitivity or anaphylaxis after FVII or IgG2 injection therapy;
3. Patients with positive FVII inhibitors or history of positive FVII inhibitors at screening;
4. Patients with severe anemia (hemoglobin < 60 g/L);
5. Patients with platelet count < 100 × 109/L;
6. Patients with abnormal liver and kidney function:

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of normal (ULN); or
   * Serum total bilirubin (TBIL) ≥ 1.5 times ULN; or
   * Serum creatinine (Cr) ≥ 1.5 times ULN or creatinine clearance < 60 mL/min calculated according to the Cockcroft-Gault formula;
7. Patients with one or more positive tests for hepatitis B virus surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus (HIV) antibody, and anti-treponema pallidum hemagglutination (TPHA)-specific antibody;
8. With the exception of hemophilia A or B, any other haemorrhagic disorders or significantly abnormal coagulation indicators (such as platelet disease, vitamin K deficiency and hypofibrinogenaemia) caused by other diseases;
9. Patients with fever, active infection and allergy (such as allergic rhinitis, allergic asthma, allergic dermatitis) within 2 weeks before the first dose;
10. Patients with severe cardiovascular and cerebrovascular diseases or thromboembolic diseases occurred within 6 months before the first dose, such as cerebral arteritis, moyamoya disease, cerebral stroke, viral myocarditis, endocarditis, endocardial fibroelastosis, severe arrhythmia, myocardial infarction, unstable angina pectoris, congestive heart failure (New York Heart Association Grade ≥ III), uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) and uncontrolled diabetes;
11. Patients receiving or planning to receive immune tolerance induction (ITI) treatment during the trial;
12. Receipt of any product containing FVII or FVIIa (plasma source or recombinant) within 24 hours before the first dose;
13. Receipt of any product containing FVIII (plasma source or recombinant) within 72 hours or 5 half-lives (whichever is longer) before the first dose or any product containing FIX (plasma source or recombinant) within 96 hours or 5 half-lives (whichever is longer) before the first dose;
14. Patients who have used any anticoagulants, antifibrinolytic agents, and chemical drugs, biological products or traditional Chinese medicines affecting platelet function within 1 week before the first dose, including non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin;
15. Patients who have received emicizumab within 6 months before the first dose;
16. Patients who have received immunomodulators (such as gamma globulin, interferon-alpha and prednisone > 10 mg/d [and > 7 days] or similar drugs, except antiretroviral drugs) within 2 weeks before the first dose;
17. Patients who have received whole blood or plasma therapy within 2 weeks before the first dose;
18. Received vaccination within 4 weeks before the first dose or planned vaccination during the PK study;
19. Patients who underwent major surgical operations (e.g. orthopedic surgery, abdominal surgery) within 1 month before the first dose, or plan to undergo surgery during the study period;
20. Patients who enrolled in other clinical trials within 1 month before the first dose;
21. Patients with a history of drug abuse or alcoholism;
22. Patients suffering from mental illness or obvious mental disorders, or incapacity or cognitive inability due to other causes;
23. Patients who have fertility plan or sperm donation plan during the whole trial period and within 3 months after administration, or are unwilling to take effective physical contraception measures (such as condom, diaphragm, intrauterine device);
24. Patients who have clinically significant diseases or other reasons that, in the opinion of the investigator, make participation in the clinical trial inappropriate (e.g., patients who cannot benefit from the clinical trial);
25. Subjects who, in the opinion of the investigator, have poor compliance that are not evaluable for efficacy or are expected to have a low likelihood of completing the intended course and follow-up.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 to Day 6
  According to the detected FVII activity of SS109 and NovoSeven®, the peak activity (Cmax)
Four-level rating scale to assess hemostasis | Day 7 to Day 96
  Hemostasis 12 h after on-demand treatment. For each new blood event, on-demand treatment should be conducted within 15min before each administration after the first dose
  The hemostatic effect of pain and bleeding symptoms/signs observed and recorded after the last treatment was evaluated according to a four-level scoring scale.
  If clinically effective (rated as "excellent" or "good") is achieved, the evaluation is discontinued.
Tmax | Day 1 to Day 6
  According to the detected FVII activity of SS109 and NovoSeven®,time to peak concentration (Tmax),
AUC0-t | Day 1 to Day 6
  area under the concentration-time curve from time 0 to the last quantifiable time point (AUC0-t) will be calculated

SECONDARY OUTCOMES:
Efficacy of hemostasis before each dose (except first dose) after treatment of all bleeding events | Day 7 to Day 96
  On-demand treatment Percentage rated "good" or "very good" before each dose after the first dose of on-demand treatmen
Time to "good" or "excellent" evaluation after treatment for all hemorrhage events | Day 7 to Day 96
  Time to "good" or "excellent" evaluation after treatment for all hemorrhage events
Evaluate the incidence of AE/SAE/AESI | Day 1 to Day 96
  Safety Measures
Incidence of positivity for FVII inhibitors | Day 1 to Day 96
  Immunogenicity Measure
anti-drug antibodies (ADAs) | Day 1 to Day 96
  Immunogenicity Measures
CHO host cell antibodies | Day 1 to Day 96
  Immunogenicity Measure

OTHER OUTCOMES:
AUC0-inf | Day 1 to Day 6
  If data allows, the area under the concentration-time curve from time 0 to infinity (AUC0-inf)
(λz | Day 1 to Day 6
  clearance (CL), elimination rate constant (λz)
t1/2 | Day 1 to Day 6
  elimination half-life
Vd | Day 1 to Day 6
  volume of distribution (Vd)
AUC_%Extrap | Day 1 to Day 6
  extrapolated percentage of area under the concentration-time curve (%) (AUC_%Extrap)
MRT | Day 1 to Day 6
  mean residence time

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - Jiangxi Provincial People's Hospital, Nanchang
  - Yangping Song, Shanxi
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin
  - Xi'an Central Hospital, Xi'an
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Provincial Cancer Hospital, Zhengzhou